CLINICAL TRIAL: NCT00613041
Title: Pilot Study: 3-D Reconstruction of CT Scan Images in the Evaluation of Non-Specific Pulmonary Nodules
Brief Title: 3-D Reconstruction of CT Scan Images in the Evaluation of Non-Specific Pulmonary Nodules
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-039
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Undiagnosed Pulmonary Nodules; Lung Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients with one or more pulmonary nodules 5-15 mm in diameter.
  Interventions: Procedure: CT Scan

INTERVENTIONS:
Procedure: CT Scan — All patients will undergo serial CT scans after 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months as is standard care. Nodules are to be scanned at 2.5mm collimation / 1.25 mm reconstruction. This resolution is necessary for volume measurements of nodules less than 1cm in diameter.

SUMMARY:
In recent years, more and more people are having lung CT scans performed to screen for various cancers. Many of them have small abnormalities detected, called "nodules", which - for a variety of reasons - doctors are unable to biopsy. As a result, many patients have their CT scans repeated on a regular basis to see if their nodules grow. This process can last several years.

Many patients experience significant anxiety during this process, when they are aware of a spot in the lung, but are not told any specific cause.

Researchers at Memorial Sloan-Kettering have developed a new way to look at lung nodules in three dimensions. The purpose of this project is to see if any change in the nodules can be detected sooner by this method than by traditional CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Referral to the pulmonary or thoracic surgery service for undiagnosed pulmonary nodules.
* History of smoking exceeding 10 pack-years (pack year defined as number of packs of cigarettes per day multiplied by the number of years smoked).
* Age >18
* Nodule size 5 to 15 mm in diameter.

Exclusion Criteria:

* Clinical indication for immediate biopsy via bronchoscopy, fine needle aspiration, or video-assisted thoracoscopic Surgery (VATS)
* Active lung cancer or metastasis to the lung.
* Contraindication to needle biopsy.
* Pneumonectomy
* Need for supplemental oxygen.
* Radiation pneumonitis
* Interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet eligibility criteria will be recruited from the services that comprise the Thoracic Disease Management Team (DMT), specifically the Divisions of Pulmonary Medicine and Thoracic Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2003-04; Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
To collect preliminary data regarding the comparative sensitivity and specificity of conventional CT scan and three-dimensional CT for detecting the growth of nonspecific pulmonary nodules. | conclusion of the study

SECONDARY OUTCOMES:
To determine three-dimensional characteristics of pulmonary nodules which may discriminate between benign and malignant diseases. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Feinstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org